CLINICAL TRIAL: NCT03511196
Title: A Phase 1b Study of Adaptive Androgen Deprivation Therapy for State IV Castration Sensitive Prostate Cancer
Brief Title: Intermittent Androgen Deprivation Therapy for Stage IV Castration Sensitive Prostate Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19367
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Stage IV Prostate Cancer; Advanced Prostate Cancer; Adenocarcinoma of the Prostate
Keywords: stage IV castration sensitive prostate cancer; advanced castration sensitive prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; abiraterone; Standard of Care; Abiraterone Acetate; Prednisone; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adaptive ADT+ Standard of Care (Experimental): Participants will undergo 12-16 weeks of GnRH analog, along with 8-12 weeks of combinational therapy with GnRH analog and abiraterone plus prednisone. 14 participants who achieve >75% PSA decline after the run-in period will be enrolled. GnRH analog and abiraterone will be stopped after study enrollment. PSA and testosterone level will be measured every 4 weeks during the run-in period, then every 6 weeks after study enrollment. Imaging studies with CT and bone scan will be performed at the time of study enrollment and these will be considered baseline scans. Study treatment will be restarted if participant's PSA reaches 2 fold or higher of his baseline PSA. Selection of treatment will be based on participant's testosterone level.
  Interventions: Drug: Adaptive Androgen Deprivation Therapy (ADT); Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: Adaptive Androgen Deprivation Therapy (ADT) — ADT with Leuprolide, Goserelin, or Triptorelin, as GnRH agonist, every 4 weeks as outlined in study arm description.
  Other Names: GnRH agonist
Drug: Abiraterone — Prednisone 5 mg once a day with food.
  Other Names: Standard of Care; Zytiga
Drug: Prednisone — Abiraterone 1000 mg daily with empty stomach.
  Other Names: Standard of Care; Glucocorticoid

SUMMARY:
Adaptive Androgen Deprivation Therapy (ADT) plus Standard of Care. The purpose of this study is to develop adaptive therapy for high risk metastatic castration sensitive prostate cancer (mCSPC).

DETAILED DESCRIPTION:
Investigators proposed this pilot feasibility study to use prostate specific antigen (PSA) response and testosterone level to guide the treatment with androgen deprivation therapy (ADT) [Leuprolide, Goserelin, and Triptorelin are the most commonly used GnRH agonists for ADT] and/or abiraterone plus prednisone. Adaptive therapy is a program of chemotherapy where the type and dosage of drug changes in an attempt to kill more of the cancer.

Abiraterone acetate with prednisone is a standard of care treatment for mCRPC (metastatic castration resistant prostate cancer). It works by interrupting the male hormone (androgen) making process in the testes, adrenal glands, and tumors. This helps to prevent the growth of tumors that need these hormones to grow.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* >75% prostate specific antigen (PSA) decline after 12 to 16 weeks of run in period with Gonadotropin-releasing Hormone (GnRH) analog abiraterone plus prednisone.
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-1
* Adequate organ function Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) must be < 2.5 x upper limit of normal (ULN), total bilirubin less than 1.5 X ULN, estimated creatinine clearance must be >40 mL/min, absolute neutrophil count (ANC) > 1500/l, hemoglobin above 9 g/dl, platelet count > 100,000/l
* Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections or major surgery within 28 days prior to study enrollment
* Ability to give written informed consent

Exclusion Criteria:

* Prior GnRH analog with GnRH analogue for non-metastatic prostate cancer within 12 months prior to study enrollment or >3 months of GnRH analog in the metastatic setting
* Prior treatments with TAK-700/Orteronel, ketoconazole, apalutamide or enzalutamide.
* Documented central nervous system metastases or liver metastasis
* Prior surgical castration
* Requiring opioids for cancer related pain.
* Treatment with any investigational compound within 30 days prior to the first dose of study drugs
* Diagnosis or treatment for another systemic malignancy within 2 years before the first dose of study drugs, or previously diagnosed with another malignancy & have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Uncontrolled hypertension despite appropriate medical therapy (blood pressure of greater than 160 mmHg systolic and 90 mmHg diastolic at 2 separate measurements no more than 60 minutes apart during the Screening period). Note: Patients may be rescreened after adjustments of antihypertensive medications
* Unstable symptomatic ischemic heart disease, ongoing arrhythmias of Grade > 2 (NCI CTCAE, version 5), New York Association Class III or IV heart failure
* Known human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C not contained with anti-viral therapy, life threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in investigator's opinion, potentially interfere with participation in this study.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of study drugs, including difficulty swallowing tables.
* Delayed healing of wounds, ulcers, and/or bone fractures
* Inability to comply with protocol requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Participant Retention | 12 months from participant's first dose of ADT
  Percentage of participants who remain on study at month 12. The study will be terminated early if 2 or more of the first 6 enrolled subjects discontinued study due to cancer progression within a year of study enrollment.

SECONDARY OUTCOMES:
Median Time to Progression From the First Dose of Androgen Deprivation Therapy (ADT) | 12 months from participant's first dose of ADT
  Median time to prostate specific antigen (PSA) progression while on androgen deprivation therapy (ADT), abiraterone and prednisone. Progression is per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and the Prostate Cancer Clinical Trials Working Group 3 (PCWG3).
Median Time to Radiographic Progression From the First Dose of ADT | 12 months from participant's first dose of ADT
  Median time to radiographic progression while on ADT, abiraterone and prednisone. Progression is per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and the Prostate Cancer Clinical Trials Working Group 3 (PCWG3).

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Result] Zhang J, Gallaher J, Cunningham JJ, Choi JW, Ionescu F, Chatwal MS, Jain R, Kim Y, Wang L, Brown JS, Anderson AR, Gatenby RA. A Phase 1b Adaptive Androgen Deprivation Therapy Trial in Metastatic Castration Sensitive Prostate Cancer. Cancers (Basel). 2022 Oct 25;14(21):5225. doi: 10.3390/cancers14215225. PMID 36358643